CLINICAL TRIAL: NCT04755686
Title: Effects of Fast-tracking Hip Fracture Patients in Geriatric Medicine Wards on Complication Incidence and Time of Hospitalization
Brief Title: Effects of Fast-tracking Geriatric Hip Fracture Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mattias Lorentzon, Associate Professor, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: dnr 154-13
Record Dates: First submitted 2013-06-10; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Hip Fracture
Keywords: hip fracture; fast-tracking; complications
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast-tracking at geriatric medicine ward (Experimental): Fast-tracking hip fracture patients at geriatric medicine ward. The goal is to optimize the medical care of older hip fracture patients at a geriatric ward and to shorten the time to operation.
  Interventions: Procedure: Fast-tracking
- Regular admission (No Intervention): Regular admission and care of hip fracture patients at the emergency room prior to surgery.

INTERVENTIONS:
Procedure: Fast-tracking
  Arms: Fast-tracking at geriatric medicine ward

SUMMARY:
The purpose of this study is to determine whether fast-tracking hip fracture patients to geriatric medicine wards, as opposed to standard care at the emergency room, results in less complications and shorter hospitalization for the patients.

DETAILED DESCRIPTION:
Each year about 18000 persons in Sweden suffer from a hip fracture. These people are often among the oldest and have many complicating diseases. The one-year mortality after hip fracture is 20%. Due to the complexity including many comorbidities in these patients, it is of great value that the care of these patients is optimal.

Today, most of the patients with suspected hip fracture in the catchment area of Sahlgrenska University hospital, Gothenburg, are transported directly to the radiology unit. Thereafter, the patient waits in the emergency room (ER) for an othopedic examination before being admitted to primarily a geriatric medicine ward where they wait for the operation. The average waiting time in the ER is today around four hours. The current scientific evidence for fast-tracking hipfracture patients is limited. The aim of our randomized controlled trial is to determine the effect of fast-tracking hip fracture patients at geraitric medicine wards compared to standard care regarding complication rate (primary endpoint), lenght of hospital stay and time to operation (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* patients with low energy trauma with pain at the hip and/or groin AND
* respiratory frequency: 8-25/minute AND
* saturation: 90% or higher on air AND
* pulse: 50-119 beats per minute AND
* systolic blood pressure: >90 mmHg AND
* level of consciousness: Reaction level scale (RLS) 1 or Glasgow Coma Scale (GCS) 14-15 AND
* plasma-glucose: 3,0-25 mmol/l

Exclusion Criteria:

We will exclude patients based on the following criteria:

* distal status affected
* suspicion of other simultaneous fracture
* suspicion of head trauma or affected consciousness
* suspicion of acute cardiac disease
* signs of acute cardiac ischemia in electrocardiogram
* generalized symtoms, except for pain in the hip

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications (composit endpoint of non-fatal major bleeding, pressure ulcer, non-fatal infections, confusion, non-fatal tromboembolic events, all-cause mortality) | at time of discharge from geriatric medicine ward, after four months and after one year

SECONDARY OUTCOMES:
Length of hospital stay, time to operation, all-cause mortality, functional ability after discharge, proportion of patients returning to former living, self assessed health status | At time of discharge from geriatric medicine ward, after four months and after one year

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Lorentzon, MD, PhD, Principal Investigator — Geriatric Medicine, Sahlgrenska University Hospital, Mölndal
Locations (1):
- Sahlgrenska University Hospital, Mölndal, Gothenburg, Sweden